CLINICAL TRIAL: NCT04074187
Title: An Open-label Multicenter Trial to Study the Efficacy and Safety of Caplacizumab in Japanese Patients With Acquired Thrombotic Thrombocytopenic Purpura
Brief Title: A Trial of Caplacizumab in Japanese Patients With Acquired Thrombotic Thrombocytopenic Purpura (aTTP)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC16297; U1111-1223-4914 (Other: UTN)
Record Dates: First submitted 2019-08-14; First posted 2019-08-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — caplacizumab; Plasma Exchange; Methylprednisolone; Prednisolone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Caplacizumab (Experimental): Eligible study participants will receive caplacizumab in addition to standard of care such as daily plasma exchange (PE) and corticosteroid treatment (mandatory), immunosuppressive treatment (if needed)
  Interventions: Drug: Caplacizumab (ALX-0081); Drug: Plasma exchange (PE); Drug: Corticosteroid treatment (Methylprednisolone or prednisolone); Drug: Immunosuppressive treatment (eg, rituximab)

INTERVENTIONS:
Drug: Caplacizumab (ALX-0081) — Pharmaceutical form:Lyophilized powder for solution for injection Route of administration: IV (first dose), SC (all subsequent doses)
Drug: Plasma exchange (PE) — Pharmaceutical form:Plasma (e.g. fresh frozen plasma) Route of administration: Plasma exchange
Drug: Corticosteroid treatment (Methylprednisolone or prednisolone) — Pharmaceutical form:Solution for injection or Tablet Route of administration: IV or Oral
Drug: Immunosuppressive treatment (eg, rituximab) — Pharmaceutical form:Solution for injection (depending on product) Route of administration: IV (depending on product)

SUMMARY:
Primary Objective:

To evaluate the effect of caplacizumab on prevention of recurrence of aTTP (proportion of participants with a recurrence of aTTP) during the overall study period.

Secondary Objectives:

* To evaluate effect of caplacizumab on

  * prevention of recurrence of TTP (the number of recurrences of TTP) during overall study period.
  * a composite endpoint consisting of aTTP-related mortality, recurrence of aTTP and major thromboembolic events during study drug treatment
  * restoring platelet counts as a measure of prevention of further microvascular thrombosis
  * refractory disease
  * biomarkers of organ damage: LDH, cardiac troponin I, serum creatinine
  * plasma exchange (PE) parameters (days of PE and volume of plasma used), days in intensive care unit, days in hospital
  * cognitive status of Japanese patients
* To evaluate safety profile of caplacizumab in Japanese patients
* To evaluate effect of caplacizumab on pharmacodynamic (PD) markers in Japanese patients
* To evaluate pharmacokinetic (PK) profile of caplacizumab in Japanese patients
* To evaluate immunogenicity of caplacizumab in Japanese patients

DETAILED DESCRIPTION:
Study duration per participant is approximately 2 months up to approximately 6 months in case of treatment extension and recurrence during the study drug treatment period.

ELIGIBILITY:
Inclusion criteria :

* Japanese participant must be 18 years or older at the time of signing the informed consent.
* Participants who have a clinical diagnosis of aTTP (initial or recurrent), which includes thrombocytopenia (defined as platelet count <100,000/µL), microangiopathic hemolytic anemia as evidenced by red blood cell fragmentation (eg, presence of schistocytes), and increased levels of LDH
* Participants who require initiation of daily PE treatment and have received a maximum of 1 PE treatment prior to enrollment in the study
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Capable of giving signed informed consent

Exclusion criteria:

* Platelet count ≥100,000/µL,
* Serum creatinine level > 2.3mg/dL in case platelet count is > 30,000µL
* Known other causes of thrombocytopenia
* Congenital TTP
* Clinically significant active bleeding or high risk of bleeding
* Malignant arterial hypertension
* Known chronic treatment with anticoagulant treatment that cannot be stopped
* Participants who were previously enrolled in a clinical study with caplacizumab and received caplacizumab or for whom the assigned treatment arm is unknown
* Participants currently or less than 28 days prior to enrollment in this study, enrolled in a clinical study with another investigational drug or device
* Clinical condition other than that associated with TTP, with life expectancy < 6 months, such as end-stage malignancy
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a recurrence of acquired thrombotic thrombocytopenic purpura (aTTP) | Approximately 2 months up to approximately 6 months
  Proportion of participants with a recurrence of aTTP during the overall study period. The success criterion for this study is proportion of evaluable participants (per-protocol population) with a recurrence of aTTP during the overall study period to be 20% or less.

SECONDARY OUTCOMES:
Number of recurrences of TTP | Approximately 2 months up to approximately 6 months
  Number of recurrences of TTP during study drug treatment (including extensions) and follow-up, as well as during overall study period.
Proportion of participants with composite endpoint consisting of aTTP-related mortality, recurrence of aTTP and major thromboembolic events | Approximately 2 months up to approximately 6 months
  Proportion of participants with TTP-related death, a recurrence of TTP, or at least one treatmentemergent major thromboembolic event (eg, myocardial infarction, cerebrovascular accident, pulmonary embolism or deep venous thrombosis [DVT]) during the overall treatment period (including extensions).
Time to platelet count response | Approximately 2 months up to approximately 6 months
  Time to platelet count response, defined as initial platelet count ≥150,000/μL with subsequent stop of daily plasma exchange (PE) within 5 days.
Proportion of participant who have a platelet count ≥150,000/μL | Approximately 2 months up to approximately 6 months
  Proportion of participant who have a platelet count ≥150,000/μL on Day 1, 2, 3, 4, 5 and Day 10 and end of study drug treatment (ie, last weekly visit during the overall treatment period).
Proportion of participants with refractory TTP | Approximately 2 months up to approximately 6 months
  Proportion of participant with refractory TTP, defined as persistent thrombocytopenia, lack of sustained platelet count increment or platelet counts <50,000/μL and persistently elevated LDH (>1.5 x upper limit of normal [ULN]) despite 5 PEs and steroid treatment.
Time to normalization of 3 organ damage marker levels | Approximately 2 months up to approximately 6 months
  Time to normalization of all 3 of the following organ damage marker levels: Time to LDH ≤ 1 x ULN, and cTnI ≤ 1 x ULN, and serum creatinine ≤ 1 x ULN and time to individual organ damage marker level.
Time to stop of daily plasma exchnage (PE) | Approximately 2 months up to approximately 6 months
  Time to stop of daily PE
Number of days to plasma exchange | Approximately 2 months up to approximately 6 months
  The endpoint will be assessed in 4 time periods: daily PE period (the first daily PE period only), overall treatment period, follow-up period (of 4 weeks after stop of study drug treatment), and overall study period
Total volume of plasma | Approximately 2 months up to approximately 6 months
  The endpoint will be assessed in 4 time periods: daily PE period (the first daily PE period only), overall treatment period, follow-up period (of 4 weeks after stop of study drug treatment), and overall study period
Number of days in ICU and in hospital | Approximately 2 months up to approximately 6 months
  Number of days in ICU and in hospital in 4 time periods: daily PE period (the first daily PE period only), overall treatment period, in the Follow-up period (of 4 weeks after stop of study drug treatment) and overall study period.
Change from baseline in the standardized mini mental state exam (SMMSE) total score | Approximately 2 months up to approximately 6 months
  Change from baseline in SMMSE total score on Day 1, (Day 2, 3, 4 as optional) and Day 5 of daily Plasma Exchange (PE) period, and Weeks 1 and 5 of the 30-day postdaily PE period, and the first (7 days after last dosing) and final follow-up (28 days after last dosing) visit.
Proportion of participants with at least one treatment emergent thromboembolic event | Approximately 2 months up to approximately 6 months
  The treatment-emergent major thromboembolic event (eg, myocardial infarction, cerebrovascular accident, pulmonary embolism or deep venous thrombosis [DVT]) during the overall treatment period (including extensions) will be evaluated.
Number of patients with treatment emergent adverse events | Approximately 2 months up to approximately 6 months
  Number of Patients with treatment emergent Adverse events (AEs) and serious adverse events (SAEs) and bleeding events
Pharmacodynamic (PD) markers | Approximately 2 months up to approximately 6 months
  PD parameters: von Willebrand factor antigen(vWF:Ag), coagulation factor VIII clotting activity (FVIII:C), von Willebrand factor ristocetin cofactor activity (vWF:RICO)
Pharmacokineticks: plasma concentration | Approximately 2 months up to approximately 6 months
  Total caplacizumab plasma concentrations
Immunogenicity of caplacizumab | Approximately 2 months up to approximately 6 months
  Anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (12):
- Japan (12):
  - Investigational Site Number 3920009, Iruma-Gun
  - Investigational Site Number 3920014, Kanazawa
  - Investigational Site Number 3920007, Kashihara-shi
  - Investigational Site Number 3920013, Kawasaki-Shi
  - Investigational Site Number 3920001, Kitakyushu-Shi
  - Investigational Site Number 3920002, Kumamoto
  - Investigational Site Number 3920003, Kurashiki-Shi
  - Investigational Site Number 3920010, Kyoto
  - Investigational Site Number 3920005, Maebashi
  - Investigational Site Number 3920015, Nagoya
  - Investigational Site Number 3920011, Osaka
  - Investigational Site Number 3920006, Sendai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Miyakawa Y, Imada K, Ichikawa S, Uchiyama H, Ueda Y, Yonezawa A, Fujitani S, Ogawa Y, Matsushita T, Asakura H, Nishio K, Suzuki K, Hashimoto Y, Murakami H, Tahara S, Tanaka T, Matsumoto M. The efficacy and safety of caplacizumab in Japanese patients with immune-mediated thrombotic thrombocytopenic purpura: an open-label phase 2/3 study. Int J Hematol. 2023 Mar;117(3):366-377. doi: 10.1007/s12185-022-03495-6. Epub 2022 Nov 24. PMID 36427162
- [Derived] Imada K, Miyakawa Y, Ichikawa S, Uchiyama H, Ueda Y, Hashimoto Y, Nishimi M, Tsukamoto M, Tahara S, Matsumoto M. Frontline use of rituximab may prevent ADAMTS13 inhibitor boosting during caplacizumab treatment in patients with iTTP: post hoc analysis of a phase 2/3 study in Japan. Thromb J. 2024 Aug 2;22(1):72. doi: 10.1186/s12959-024-00642-3. PMID 39095866
- See also: EFC16297 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25244&tenant=MT_SNY_9011